CLINICAL TRIAL: NCT05602350
Title: Testing Response Bias on Sensitive Topics in Self- Versus Enumerator-administered Surveys
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chicago (Other)
Collaborators: Innovations for Poverty Action (Other)
Responsible Party: Principal Investigator, Christopher Blattman, Ramalee E. Pearson Professor of Global Conflict Studies, University of Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB19-1212
Record Dates: First submitted 2022-09-23; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Bias, Implicit
MeSH Terms: conditions — Bias, Implicit

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Survey respondents will self-administer three survey sections in a tablet: (1) antisocial behaviors, (2) depression symptoms, and (3) anxiety symptoms
  Interventions: Behavioral: Self-administered survey
- Control (Placebo Comparator): Survey respondents will have the survey questions on the three sections administered by an enumerator
  Interventions: Behavioral: Enumerator-administered survey

INTERVENTIONS:
Behavioral: Self-administered survey — Subjects will self-administer questionnaire sections on sensitive topics: (1) antisocial behaviors, (2) symptoms of depression, and (3) symptoms of anxiety.
  Arms: Treatment
Behavioral: Enumerator-administered survey — Subjects will have enumerator-administered questionnaire sections on sensitive topics: (1) antisocial behaviors, (2) symptoms of depression, and (3) symptoms of anxiety.
  Arms: Control

SUMMARY:
Within a survey of adolescent males in Medellin schools (mainly 13-year old boys) the researchers are randomizing whether survey respondents answer sensitive questions themselves or are asked the questions by an enumerator. Questions are of three main varieties: (1) antisocial behaviors, (2) symptoms of depression, and (3) symptoms of anxiety.

ELIGIBILITY:
Inclusion Criteria:

* All male students in seventh grade in a sample of public schools are eligible. The sample corresponds to a representative sample of public schools (we aim at 90 schools)

Exclusion Criteria:

* Female students or students not in seventh grade

Ages: 9 Years to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7500 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
The main outcome is the mean difference in survey responses for an average of the three indexes being measured | Through study completion, an average of 1 year
  Three survey sections are being tested: (1) antisocial behaviors, (2) depression symptoms, and (3) anxiety symptoms. Each section can be summarized by a single index of survey questions in that section--indexes of antisocial behavior, depression and anxiety. To reduce the number of hypotheses tested, the researchers plan to test the difference by treatment status for an average of these three indexes. The researchers also plan to test the mean difference by treatment status for each of the three indexes, and will report regular standard errors as well as standard errors corrected for three comparisons.

CONTACTS AND LOCATIONS:
Locations (1):
- Innovations for Poverty Action, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No